CLINICAL TRIAL: NCT03198390
Title: Linking Epidermal Barrier Function With Anti-Oxidant Defense Mechanisms in Skin Conditions
Status: Terminated | Type: Observational
Why Stopped: Investigator left university
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 1705434989
Record Dates: First submitted 2017-06-13; First posted 2017-06-26 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Atopic Dermatitis; Hidradenitis Suppurativa; Contact Dermatitis; Psoriasis
MeSH Terms: conditions — Dermatitis, Atopic; Hidradenitis Suppurativa; Dermatitis, Contact; Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with chronic skin conditions: Subjects with chronic skin conditions including but not limited to atopic dermatitis, contact dermatitis, hidradenitis suppurativa, and psoriasis
- Healthy subjects

SUMMARY:
Investigators will sample the skin and blood of patients with chronic skin conditions (including but not limited to atopic dermatitis (AD), contact dermatitis, hidradenitis suppurativa (HS), and psoriasis) to study the expression of anti-oxidative enzymes, skin barrier proteins and inflammatory molecules. In patients with atopic dermatitis, investigators will also measure skin barrier function using noninvasive devices. These results will be correlated with the disease severity in atopic dermatitis patients.

DETAILED DESCRIPTION:
Up to 300 subjects with chronic skin conditions (including but not limited to atopic dermatitis (AD), contact dermatitis, hidradenitis suppurativa (HS), and psoriasis) and 100 healthy subjects meeting the inclusion criteria will be enrolled. Medical records will be reviewed pertaining to the subject's diagnosed chronic skin condition and specific therapeutic interventions.

For atopic dermatitis subjects, AD severity will be assessed using Eczema Area and Severity Index (EASI). Study sites will be chosen by the investigator. One lesional and one nonlesional site on the trunk, upper, or lower extremities will be selected. Digital photos of the study skin site(s) will be taken. Skin barrier function indices (transepidermal water loss, pH, sebum and hydration levels) of an active lesion and adjacent nonlesional skin will be measured using noninvasive skin barrier measurement devices.

For subjects with other chronic skin conditions such as contact dermatitis, HS or psoriasis, photos of the selected study sites will be taken. No skin barrier measurements will be performed.

For all subjects, two 3mm punch biopsies will be performed over the selected skin sites. One biopsy will be performed over an active lesion and another on adjacent nonlesional skin. Tissue will be sent out for immunohistochemical staining to study the expression anti-oxidant biomarkers. Five mL of peripheral venous blood will be collected for immunoassay to measure the level inflammatory cytokines.

For healthy subjects, digital photo of the study skin site(s) over either the trunk, upper, or lower extremities will be taken. Skin barrier function indices (transepidermal water loss, pH, sebum and hydration levels) of skin be measured using noninvasive skin barrier measurement devices. One 3mm punch biopsy will be performed over the same skin site that skin barrier measurements were performed. Tissue will be sent out for immunohistochemical staining to study the expression anti-oxidant biomarkers. Five mL of peripheral venous blood will be collected for immunoassay to measure the level inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

Male and female 18 to 99 years of age. Chronic skin conditions (including but not limited to atopic dermatitis, contact dermatitis, hidradenitis suppurativa, and psoriasis) with at least one active skin lesion Healthy skin (defined no clinical evidence or diagnosis of inflammatory skin conditions)

Exclusion Criteria:

Subjects who are unable to comply with study procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female, from 18 to 99 years of age.Adult subjects must be able to comprehend and read the English language. Subjects diagnosed with chronic skin conditions or with healthy skin defined as without clinical evidence or diagnosis of inflammatory skin conditions. Subjects with chronic skin conditions must have at least one active skin lesion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Skin barrier function | 1 hour
  Transepidermal water loss (TEWL) status will be measured using hand-held, noninvasive, skin barrier measuring device (Tewameter).
Skin barrier function | 1 hour
  Stratum corneum hydration status will be measured using hand-held, noninvasive, skin barrier measuring device (Moisturemeter/Corneometer)
Skin pH | 1 hour
  Skin pH will be measured using a pH meter.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona - Banner University Medicine Dermatology, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No